CLINICAL TRIAL: NCT02056457
Title: Parents and Children Together
Brief Title: An Evaluation of Selected Responsible Fatherhood and Healthy Marriage Programs: Parents and Children Together
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: MPR06997
Record Dates: First submitted 2014-01-31; First posted 2014-02-06 (Estimated); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Responsible Fatherhood; Healthy Marriage
Keywords: Responsible fatherhood; Healthy marriage; Healthy relationships; Parenting; Economic self-sufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Responsible fatherhood or healthy marriage (Experimental)
  Interventions: Behavioral: Responsible Fatherhood or Healthy Marriage Program
- Control (Experimental)
  Interventions: Behavioral: Other services in the community

INTERVENTIONS:
Behavioral: Responsible Fatherhood or Healthy Marriage Program — RF grantees funded by the most recent re-authorization of the program must offer services in each of three categories: (1) healthy marriage; (2) responsible parenting; and (3) economic stability. HM grantees must provide one or more of eight allowable activities, which include marriage and relationship skills programs, mentoring, divorce reduction programs, and education in high schools on the value of marriage, relationships skills, and budgeting.
  Arms: Responsible fatherhood or healthy marriage
Behavioral: Other services in the community — RF grantees funded by the most recent re-authorization of the program must offer services in each of three categories: (1) healthy marriage; (2) responsible parenting; and (3) economic stability. HM grantees must provide one or more of eight allowable activities, which include marriage and relationship skills programs, mentoring, divorce reduction programs, and education in high schools on the value of marriage, relationships skills, and budgeting.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the effectiveness of selected healthy marriage (HM) and responsible fatherhood (RF) grant programs, authorized by by the Claims Resolution Act of 2010. The programs are intended to improve the well-being of parents and families in domains such as economic self-sufficiency, parenting, and healthy relationships.

DETAILED DESCRIPTION:
Since 2006, Congress has provided funding for grants to provide healthy marriage and responsible fatherhood services to help interested couples and fathers enhance or improve adult and parent-child relationships and meet other objectives. The Administration for Children and Families (ACF), within the Department of Health and Human Services (HHS), oversees these grants and provides supports to assist grantees to meet their goals and objectives. To learn about the implementation and effects of these programs, ACF awarded a contract in 2011 to Mathematica Policy Research, Inc. to conduct the Parents and Children Together (PACT) evaluation. The evaluation includes separate impact and process studies for responsible fatherhood and healthy marriage programs.

Individuals who are eligible for the programs and agree to be in the study are randomly assigned to either a program group or a control group. Program group members are offered program services; control group members are not offered those services but are able to receive other services available in the community. The impact studies will examine whether the programs improve outcomes for fathers, mothers, families, and children in the program group compared to outcomes of those in the control group. Members of both program and control groups are surveyed twice: before they are randomly assigned and 12 months later. At the 12-month follow-up, both groups will be asked to complete a telephone survey. The survey will cover a range of questions related to adult relationships and interactions, parent-child interactions and economic stability. Corresponding process studies will examine multiple aspects of the implementation and operation of the programs. Information for the process studies will be obtained through: interviews with program and partner organization managers and staff; observations of program operations; from focus groups with program participants and non-participants; and from data from each grantee's management information system.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the PACT HM Evaluation, the applicant must be part of a couple (as defined by the couple) in which both couple members are applying to the program and that:

  1. Both members of the couple are eligible for the program
  2. Both members of the couple are 18 years of age or older
  3. One member of the couple is female and the other male
  4. At least one member of the couple is an expectant parent or a parent of a biological or adoptive child who is living with him or her (That is the children do not need to be children in common and they need to be living with only one parent)
* To be eligible for the PACT RF evaluation, the individual must:

  1. Be male
  2. Be 18 years or older
  3. Have a living biological or adopted child or is expecting a child

Exclusion Criteria:

* Does not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2012-12; Primary Completion 2015-04 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
In-person contact with child(ren) in past month | 12 months
Earnings in past year | 12 months
Co-parenting teamwork | 12 months
  Agreement with whether father and mother work well together as parents

CONTACTS AND LOCATIONS:
Overall Officials: Sheena McConnell, Ph.D., Study Director — Mathematica Policy Research; Robin Dion, M.A., Study Director — Mathematica Policy Research
Locations (7):
- United States (7):
  - Jewish Family and Children's Services, Sarasota, Florida
  - Goodwill/Easter Seals Minnesota, Minneapolis, Minnesota
  - Urban Ventures, Minneapolis, Minnesota
  - Connections to Success, Kansas City, Missouri
  - Fathers' Support Center, St Louis, Missouri
  - University Behavioral Associates, The Bronx, New York
  - El Paso Center for Children, El Paso, Texas